CLINICAL TRIAL: NCT02550067
Title: A Multi Center, Open-Label, Randomised Clinical Trial Comparing HIV Incidence and Contraceptive Benefits in Women Using Depot Medroxyprogesterone Acetate (DMPA), Levonorgestrel (LNG) Implant, and Copper Intrauterine Devices (IUDs)
Brief Title: The Evidence for Contraceptive Options and HIV Outcomes Trial
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: University of Washington (Other); Wits Reproductive Health and HIV Institute (Other); World Health Organization (Other); Madibeng Centre for Research (Other); Maternal Adolescent and Child Health Research (Unknown); Qhakaza Mbokodo Research Clinic (Unknown); The Aurum Institute NPC (Other); Effective Care Research Unit (Other); Emavundleni Research Centre (Unknown); Setshaba Research Centre (Unknown); University of North Carolina, Chapel Hill (Other); Family Life Association of Swaziland (Unknown); ICAP Columbia University (Unknown); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 523201
Record Dates: First submitted 2015-09-12; First posted 2015-09-15 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: HIV; Contraception
Keywords: HIV infection; DepoLevonorgestrel; Contraception; DMPA; Copper IUD; Levonorgestrel implant; IUD
MeSH Terms: conditions — HIV Infections | interventions — N,N-dimethyl-4-anisidine; Levonorgestrel; Intrauterine Devices, Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Depot medroxyprogesterone acetate (DMPA) (Active Comparator): Women randomized to DMPA, will receive an intramuscular injection of DMPA (medroxyprogesterone acetate sterile aqueous suspension 150 mg per 1 mL) at enrolment. Subsequent injections will be given every 3 months (i.e., at quarterly study visits) at the study site.
  Interventions: Drug: DMPA
- Levonorgestrel implant (LNG) (Active Comparator): Women randomized to implants will receive LNG implants in the arm, at enrolment from trained clinicians.
  Interventions: Drug: LNG
- Copper T380a IUD (Active Comparator): Women randomized to IUDs will receive their IUDs at enrolment. Trained providers will insert T380a copper IUDs using standard insertion techniques.
  Interventions: Drug: Copper IUD

INTERVENTIONS:
Drug: DMPA — Women randomized to DMPA, will receive an intramuscular injection of DMPA (medroxyprogesterone acetate sterile aqueous suspension 150 mg per 1 mL) at enrolment. Subsequent injections will be given every 3 months (i.e., at quarterly study visits) at the study site.
  Other Names: Depot medroxyprogesterone acetate
  Arms: Depot medroxyprogesterone acetate (DMPA)
Drug: LNG — Women randomized to implants will receive LNG implants in the arm, at enrolment from trained clinicians.
  Other Names: Levonorgestrel implant
  Arms: Levonorgestrel implant (LNG)
Drug: Copper IUD — Women randomized to IUDs will receive their IUDs at enrolment. Trained providers will insert T380a copper IUDs using standard insertion techniques.
  Other Names: Copper T380a IUD
  Arms: Copper T380a IUD

SUMMARY:
The ECHO Study is an open-label randomized clinical trial that will compare three highly effective, reversible methods of contraception (including a non-hormonal method) to evaluate whether there is a link between use of any of these methods and increased risk of acquiring HIV infection. A randomized clinical trial among about 7,800 women in four countries, ECHO will deliver evidence to support and guide individual, policy and programmatic decisions on contraception for women at risk of acquiring HIV infection.

DETAILED DESCRIPTION:
Approximately 7800 sexually active, HIV-negative women, 16-35 years old, seeking effective contraception, willing to be randomized to any of the study arms, and not desiring pregnancy for the duration of study participation will be randomly allocated to one of three study arms in a 1:1:1 ratio: depot medroxyprogesterone acetate (DMPA), levonorgestrel (LNG) implant, copper intrauterine device (IUD).

Enrollment will require an estimated 18 months and the total duration of the clinical portion of the study is estimated to be 36 months.

The primary objective is to compare the risks of HIV acquisition between women randomized to DMPA, levonorgestrel (LNG) implant, and copper IUDs. Secondary objectives are to compare: 1) pregnancy rates among women randomized to DMPA, LNG implant, and copper IUDs, 2) rates of serious adverse events among women randomized to DMPA, LNG implant, and copper IUDs, 3) rates of adverse events that lead to method discontinuation among women randomized to DMPA, LNG implant, and copper IUDs, and 4) contraceptive method continuation rates among women randomized to DMPA, LNG implant, and copper IUDs. Tertiary objectives are to evaluate: 1) whether age modifies the relationship between the three contraceptive methods and HIV acquisition, 2) whether HSV-2 status modifies the relationship between the three contraceptive methods and HIV acquisition, and 3) early HIV disease progression among sero-converters randomized to DMPA, LNG implant, and copper IUDs. Ancillary studies will assess biological mechanisms at the interface of contraceptives and markers of HIV risk.

ELIGIBILITY:
Inclusion Criteria:

* 16-35 years of age (previously pregnant 16 and 17 year olds, where permissible by national regulations and local IRB approval)
* HIV-seronegative
* Wants to use effective contraception
* Is able and willing to provide written informed consent
* Agrees to be randomized to either DMPA, LNG implant, or copper IUD
* Agrees to use assigned method for 18 months
* Agrees to follow all study requirements
* Intends to stay in the study area for the next 18 months, and willing and able to provide adequate locator information
* If has had a recent third trimester birth, is at least 6 weeks postpartum
* Is sexually active (has had vaginal sex within the last 3 months) or was pregnant within the last 3 months
* Agrees not to participate in studies of drugs or vaccines or any other clinical research study while participating in this study.

Exclusion Criteria:

* Reported medical contraindications (WHO MEC Category 3 or 4) to DMPA, LNG implant, or copper IUDs, including: recent septic abortion; suspicious unexplained vaginal bleeding; breast, cervical, uterine, or ovarian cancer; high BP or heart disease, venous thromboembolism, stroke, or diabetes; liver disease or liver tumours; use of liver enzyme inducing medications
* Is found to have pelvic tuberculosis or uterine fibroids with distortion of the uterine cavity on pelvic exam
* Has untreated mucus and purulent cervicitis on exam, untreated pelvic inflammatory disease (PID), or untreated known gonorrhea or chlamydia
* Has received a DMPA or NET-En injection in the last 6 months
* Has used an implant or an IUD in the last 6 months
* Is pregnant or intending to become pregnant in the next 18 months
* Has had a hysterectomy or sterilization
* Has previously participated in the study
* Has any condition (social or medical) which in the opinion of the investigator would make study participation unsafe or complicate data interpretation.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7830 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Compare risks of HIV acquisition between women randomized to DMPA, LNG and copper IUD | From enrollment to 18 months
  HIV infection as measured by documented HIV seroconversion occurring post-enrolment

SECONDARY OUTCOMES:
Compare pregnancy rates among women randomized to DMPA, LNG and copper IUD | From enrollment to 18 months
Compare rates of adverse events that lead to discontinuation among women randomized to DMPA, LNG and copper IUD | From enrollment to 18 months
Compare contraceptive continuation rates among women randomized to DMPA, LNG and copper IUD | From enrollment to 18 months
Compare SAEs among women randomized to DMPA, LNG and copper IUD | From enrollment to 18 months

CONTACTS AND LOCATIONS:
Locations (12):
- FLAS/ICAP Clinic 1& Clinic 2, Manzini, Eswatini
- Kisumu East Research Care and Training Program, Kisumu, Kenya
- South Africa (9):
  - Madibeng Centre for Research, Brits
  - Emavundleni Research Centre, Cape Town
  - MatCH Research Unit Commercial City, Durban
  - Effective Care Research Unit (ECRU) Frere Maternity Hospital, East London
  - Wits Reproductive Health and HIV Institute (WRHI), Johannesburg
  - Aurum Klerksdorp Gavin Churchyard Legacy Centre, Klerksdorp
  - QM ladysmith, Ladysmith
  - MatCH Research Unit Edendale, Pietermaritzburg
  - Setshaba Research Centre, Soshanguve
- University Teaching Hospital, Lusaka, Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary analysis, after deidentification, are available beginning 3 months following article publication ending after 36 months. The study protocol is available upon publication.The statistical code is available 3 months after publication from the corresponding author. Data is available for researchers who provide a methodologically sound proposal, which will be reviewed by the ECHO Management Committee. Proposals should be directed to icrc@uw.edu; to gain access, data requestors will need to sign a data access agreement and any proposal will require approval by the ECHO Management Committee.
Supporting Information: Study Protocol, ICF
Time Frame: The data are available 3 months following publication of primary analysis, for 36 months.

REFERENCES:
- [Derived] Morrison S, Batting J, Wanga V, Beesham I, Deese J, Hofmeyr GJ, Kasaro MP, Louw C, Morrison C, Mugo NR, Palanee-Phillips T, Pleaner M, Reddy K, Scoville CW, Smit J, Stringer JSA, Ahmed K, Bukusi E, Kotze P, Baeten JM; ECHO Trial Team. True and False Positive HIV Point of Care Test Results in a Prospective Multinational Study of At-Risk African Women: Implications for Large-Scale Repeat HIV Testing in HIV Prevention Programs. J Acquir Immune Defic Syndr. 2024 Dec 1;97(4):364-370. doi: 10.1097/QAI.0000000000003497. PMID 39085989
- [Derived] Hofmeyr GJ, Singata-Madliki M, Batting J, Balakrishna Y, Morroni C. Effects of depot medroxyprogesterone acetate, the copper IUD and the levonorgestrel implant on testosterone, sex hormone binding globulin and free testosterone levels: ancillary study of the ECHO randomized clinical trial. BMC Womens Health. 2024 Mar 8;24(1):167. doi: 10.1186/s12905-024-02990-8. PMID 38459552
- [Derived] Beesham I, Mansoor LE, Joseph Davey DL, Palanee-Phillips T, Smit J, Ahmed K, Selepe P, Louw C, Singata-Madliki M, Kotze P, Heffron R, Parikh UM, Wiesner L, Rees H, Baeten JM, Beksinska M. Brief Report: Quantifiable Plasma Tenofovir Among South African Women Using Daily Oral Pre-exposure Prophylaxis During the ECHO Trial. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):26-30. doi: 10.1097/QAI.0000000000003023. Epub 2022 Jun 9. PMID 35972853
- [Derived] Bunjun R, Ramla TF, Jaumdally SZ, Noel-Romas L, Ayele H, Brown BP, Gamieldien H, Harryparsad R, Dabee S, Nair G, Onono M, Palanee-Phillips T, Scoville CW, Heller KB, Baeten JM, Bosinger SE, Burgener A, Passmore JS, Jaspan H, Heffron R. Initiating Intramuscular Depot Medroxyprogesterone Acetate Increases Frequencies of Th17-like Human Immunodeficiency Virus Target Cells in the Genital Tract of Women in South Africa: A Randomized Trial. Clin Infect Dis. 2022 Nov 30;75(11):2000-2011. doi: 10.1093/cid/ciac284. PMID 35941737
- [Derived] Ryan R, Mussa A, Singtaa-Madliki M, Batting J, Balakrishna Y, Morroni C, Hofmeyr GJ. Effects of Depot Medroxyprogesterone Acetate Intramuscular Injection, Copper Intrauterine Device and Levonorgestrel Implant Contraception on Estradiol Levels: An Ancillary Study of the ECHO Randomized Trial. Front Glob Womens Health. 2022 May 20;3:887541. doi: 10.3389/fgwh.2022.887541. eCollection 2022. PMID 35669313
- [Derived] Palanee-Phillips T, Rees HV, Heller KB, Ahmed K, Batting J, Beesham I, Heffron R, Justman J, Makkan H, Mastro TD, Morrison SA, Mugo N, Nair G, Kiarie J, Philip NM, Pleaner M, Reddy K, Selepe P, Steyn PS, Scoville CW, Smit J, Thomas KK, Donnell D, Baeten JM; ECHO Trial Consortium. High HIV incidence among young women in South Africa: Data from a large prospective study. PLoS One. 2022 Jun 3;17(6):e0269317. doi: 10.1371/journal.pone.0269317. eCollection 2022. PMID 35657948
- [Derived] Tanko RF, Bunjun R, Dabee S, Jaumdally SZ, Onono M, Nair G, Palanee-Phillips T, Harryparsad R, Happel AU, Gamieldien H, Qumbelo Y, Sinkala M, Scoville CW, Heller K, Baeten JM, Bosinger SE, Burgener A, Heffron R, Jaspan HB, Passmore JAS. The Effect of Contraception on Genital Cytokines in Women Randomized to Copper Intrauterine Device, Depot Medroxyprogesterone Acetate, or Levonorgestrel Implant. J Infect Dis. 2022 Sep 13;226(5):907-919. doi: 10.1093/infdis/jiac084. PMID 35263421
- [Derived] Mugo NR, Stalter RM, Heffron R, Rees H, Scoville CW, Morrison C, Kourtis AP, Bukusi E, Beksinka M, Philip NM, Beesham I, Deese J, Edward V, Donnell D, Baeten JM; Evidence for Contraceptive Options and HIV Outcomes (ECHO) Trial Consortium. Incidence of Herpes Simplex Virus Type 2 Infection Among African Women Using Depot Medroxyprogesterone Acetate, a Copper Intrauterine Device, or a Levonorgestrel Implant for Contraception: A Nested Randomized Trial. Clin Infect Dis. 2022 Sep 10;75(4):586-595. doi: 10.1093/cid/ciab1027. PMID 34910143
- [Derived] Donnell D, Beesham I, Welch JD, Heffron R, Pleaner M, Kidoguchi L, Palanee-Phillips T, Ahmed K, Baron D, Bukusi EA, Louw C, Mastro TD, Smit J, Batting JR, Malahleha M, Bailey VC, Beksinska M, Rees H, Baeten JM; ECHO Trial Consortium. Incorporating oral PrEP into standard prevention services for South African women: a nested interrupted time-series study. Lancet HIV. 2021 Aug;8(8):e495-e501. doi: 10.1016/S2352-3018(21)00048-5. Epub 2021 Jun 11. PMID 34126052
- [Derived] Beksinska M, Issema R, Beesham I, Lalbahadur T, Thomas K, Morrison C, Hofmeyr GJ, Steyn PS, Mugo N, Palanee-Phillips T, Ahmed K, Nair G, Baeten JM, Smit J. Weight change among women using intramuscular depot medroxyprogesterone acetate, a copper intrauterine device, or a levonorgestrel implant for contraception: Findings from a randomised, multicentre, open-label trial. EClinicalMedicine. 2021 Apr 6;34:100800. doi: 10.1016/j.eclinm.2021.100800. eCollection 2021 Apr. PMID 33898953
- [Derived] Beesham I, Welch JD, Heffron R, Pleaner M, Kidoguchi L, Palanee-Phillips T, Ahmed K, Baron D, Bukusi EA, Louw C, Mastro TD, Smit J, Batting JR, Malahleha M, Bailey VC, Beksinska M, Donnell D, Baeten JM; ECHO Trial Consortium. Integrating oral PrEP delivery among African women in a large HIV endpoint-driven clinical trial. J Int AIDS Soc. 2020 May;23(5):e25491. doi: 10.1002/jia2.25491. PMID 32396700
- [Derived] Evidence for Contraceptive Options and HIV Outcomes (ECHO) Trial Consortium. HIV incidence among women using intramuscular depot medroxyprogesterone acetate, a copper intrauterine device, or a levonorgestrel implant for contraception: a randomised, multicentre, open-label trial. Lancet. 2019 Jul 27;394(10195):303-313. doi: 10.1016/S0140-6736(19)31288-7. Epub 2019 Jun 13. PMID 31204114